CLINICAL TRIAL: NCT05663710
Title: Phase 1b/2 Study of Combination 177Lu Girentuximab Plus Cabozantinib and Nivolumab in Treatment naïve Patients With Advanced Clear Cell RCC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Telix Pharmaceuticals Limited (Unknown); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0911; NCI-2022-10595 (Other: NCI-CTRP Clinical Trials Registry); CDMRP-KC210253 (Other: CDMRP-eBRAP Log Number)
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Advanced Cancer; Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Biopsy) (Experimental): Participants within 2 weeks of starting the first dose of 177Lu-girentuximab
  Interventions: Drug: 177Lu girentuximab; Drug: Nivolumab; Drug: Cabozantinib; Drug: ArabinoFuranosylGuanine [18F]F-AraG
- Cohort 2 (Biopsy) (Experimental): Participants within 2 weeks of Cycle 4
  Interventions: Drug: 177Lu girentuximab; Drug: Nivolumab; Drug: Cabozantinib; Drug: ArabinoFuranosylGuanine [18F]F-AraG
- Cohort 3 (Biopsy) (Experimental): Participants at the time of progression or at 20 months post treatment
  Interventions: Drug: 177Lu girentuximab; Drug: Nivolumab; Drug: Cabozantinib; Drug: ArabinoFuranosylGuanine [18F]F-AraG

INTERVENTIONS:
Drug: 177Lu girentuximab — Given by IV (vein)
Drug: Nivolumab — Given by IV (vein)
  Other Names: BMS-936558; Opdivo
Drug: Cabozantinib — Given by PO
  Other Names: XL-184; XL184
Drug: ArabinoFuranosylGuanine [18F]F-AraG — Given by IV (vein)

SUMMARY:
To learn if giving 177Lu girentuximab in combination with cabozantinib plus nivolumab can help to control advanced clear cell renal cell carcinoma (ccRCC).

DETAILED DESCRIPTION:
Primary Objectives:

* To determine safety of combination 177Lu girentuximab in combination with nivolumab plus cabozantinib in subjects with previously untreated ccRCC.
* To evaluate CR rate in the combination of 177Lu girentuximab with nivolumab plus cabozantinib in subjects with previously untreated ccRCC. 2. CR rate by RECIST 1.1 by investigator

Secondary Objectives:

* To evaluate ORR of 177Lu girentuximab in combination with nivolumab plus cabozantinib in subjects with previously untreated ccRCC.
* To evaluate PFS of 177Lu girentuximab in combination with nivolumab plus cabozantinib in subjects with previously untreated ccRCC.

ELIGIBILITY:
Inclusion Criteria:

1. Has the ability to understand and willingness to sign a written ICF before the performance of any study-specific procedures on this protocol and 2022-0515
2. Age ≥ 18 years
3. Has locally advanced or metastatic RCC with predominantly clear cell subtype
4. Has at least one measurable lesion as defined by RECIST version 1.1
5. Has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1
6. Has adequate organ function defined as follows:

   a. Absolute neutrophil count ≥ 1,500/µL, Hgb level ≥ 9 g/dL and platelet count (Plt) i. ≥ 100,000/µL without transfusion or growth factor support within 2 weeks prior to obtaining the hematology values at screening; b. Creatinine clearance ≥ 40 mL/min/1.73m2 c. Transaminase levels (AST/ALT) ≤ 3.0 × upper limit of normal (ULN); total bilirubin i. (TBILI) ≤ 1.5 mg/dL in the absence of Gilbert's disease
7. Women of child beariring potential must have a negative serum preganancy test within 7 days before first study drug administration
8. Female patients of child bearing potential, or a male patients with a female partner of child-bearing potential (defined as all women physiologically capable of becoming pregnant), must agree to use a highly effective method of contraception during screening, during the period of drug administration and for 120 days after stopping study drug administration. Highly effective contraception methods include the following:

   1. Total abstinence (defined as refraining from heterosexual intercourse during the entire period outlined above),
   2. Male or female sterilization, or

   Use of at least one of the following:

   Use of oral, injectable, transdermal, intravaginal, or implantable hormonal methods of contraception i. Combined estrogen and progestogen containing hormonal contraception associated with inhibition of ovulation ii. Progestogen-only hormonal contraception associated with inhibition of ovulation c. Placement of an intrauterine device or intrauterine system
9. Able to swallow oral medications
10. Able to provide tumor tissue sample (archival or recent acquisition)
11. Patients with brain metastases are eligible providing other measurable disease exists and brain lesions are controlled for one month (requiring no therapy) and are not life threatening.

Exclusion Criteria:

1. Has received treatment with any frontline systemic therapy for metastatic RCC
2. Has a history of leptomeningeal disease or spinal cord compression
3. Has a history of autoimmune disease requiring active therapy
4. Has a history of brain metastases except:

   1. Patients may be enrolled if they have treated brain metastases with no evidence of progression or hemorrhage after therapy for brain metastases (e.g. radiation therapy, surgery, radiosurgery) AND
   2. Patients may be enrolled if they do not require ongoing treatment with dexamethasone or anti-epileptic drugs
5. Has had radiation therapy for bone metastases within 2 weeks, or any other external radiation therapy (5 days or longer) to sites other than bone, within 4 weeks before administration of the first dose of study treatment. Patients with clinically relevant ongoing major complications from prior radiation therapy are not eligible.
6. Has uncontrolled or poorly controlled hypertension, as defined by a sustained blood pressure (BP) > 140/90 with or without antihypertensive treatment
7. Has had any major cardiovascular event within 6 months prior to study drug administration including but not limited to myocardial infarction, unstable angina, cerebrovascular accident, transient ischemic attack, pulmonary embolism, clinically significant ventricular arrhythmias (e.g. sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes) or New York Heart Association Class III or IV heart failure
8. Has any other clinically significant cardiac, respiratory, or other medical or psychiatric condition that might interfere with participation in the trial or interfere with the interpretation of trial results, in the opinion of the investigator or medical monitor
9. Has an active infection requiring systemic treatment
10. Is participating in another therapeutic clinical trial
11. Is receiving chronic concomitant treatment with strong CYP3A4 inducers or CYP3A4 inhibitors
12. Has manifestations of malabsorption due to prior gastrointestinal (GI) surgery or GI disease
13. Has GI disorders including those associated with a high risk of perforation or fistula formation:

    1. Tumors invading the GI-tract, active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic or biliary duct, or gastric outlet obstruction
    2. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before administration of the first dose of study treatment. Note: complete healing of an intra-abdominal abscess must be confirmed before administration of the first dose of study treatment
14. Has tumor invading or encasing any major blood vessels
15. Has other clinically significant disorders such as:

    1. Serious non-healing wound/ulcer/bone fracture
    2. Moderate to severe hepatic impairment (Child-Pugh B or C).
    3. Requirement for hemodialysis or peritoneal dialysis
    4. History of solid organ transplantation
16. Has had major surgery (e.g., GI surgery, removal or biopsy of brain metastasis) within 2 months before the first study drug administration. Complete wound healing from major surgery must have occurred 1 month before the first study drug administration and from minor surgery (e.g., simple excision, tooth extraction) at least 10 days before the first study drug administration. Patients with clinically relevant ongoing complications from prior surgery are not eligible
17. Has a prior or concomitant invasive malignancy other than RCC with the exception of adequately treated basal or squamous cell carcinoma of the skin, cervical carcinoma in situ or any other malignancy from which the patient has remained disease free for more than 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org